CLINICAL TRIAL: NCT04464499
Title: Validation Study of WITHINGS BPM Core for the Detection of Atrial Fibrillation
Acronym: Core AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A03346-51
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases
Keywords: atrial fibrillation; arrhythmia, cardiac; cardiovascular disease; heart disease; wearable electronic device; ECG; blood pressure monitor; electrocardiography
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- atrial fibrillation (AF): Patients diagnosed with AF during reference ECG
  Interventions: Diagnostic Test: ECG measurement
- sinus rhythm (SR): Patients diagnosed with SR during reference ECG
  Interventions: Diagnostic Test: ECG measurement

INTERVENTIONS:
Diagnostic Test: ECG measurement — Simultaneous recording of a single-lead ECG signal with the Withings BPM Core and ECG signal for the reference 12-lead ECG

SUMMARY:
The proposed clinical study aims to validate the diagnostic performance, compared to a reference ECG, of the electrocardiographic function of the BPM Core developed by Withings for the automatic identification of atrial fibrillation (AF).

DETAILED DESCRIPTION:
BPM Core is a blood-pressure monitor with an build-in single-channel electrocardiogram similar to a lead I.

Primary objective:

The primary objective is to demonstrate that Withings BPM Core has acceptable sensitivity and specificity in the automatic identification of AF and SR in comparison with a gold-standard diagnosis from a 12-lead ECG by board certified cardiologists.

The algorithm classifies the device signals into four categories: normal sinus rhythm (RSN), AF, arrhythmia other than AF, or non-interpretable. The latter category includes signals of insufficient quality to be interpreted with confidence.

This classification will be compared to the diagnosis made by three independent, blinded cardiologists based on a 12-lead ECG. The final diagnosis retained will be decided by majority with adjudication by a consensus of 3 to 6 cardiologists. The sensitivity and specificity of the device will then be estimated.

Secondary objectives:

The first secondary objective is to assess the quality of tracings of the BPM Core armband thanks to a qualitative and quantitative comparison between BPM Core tracings and reference ECG ones, based on clinical evaluation criteria.

Firstly, three independent cardiologists who have not performed or read the reference ECG and do not know the patient's clinical files will make a diagnosis from the recordings from the BPM Core. There will be a majority vote to select the diagnosis. The cases where the three readers reached three different diagnosis will be reviewed by a panel of 3 to 6 board certified cardiologists who will decide by consensus. Sensitivity and specificity will be calculated relative to the reference ECG.

Secondly, quantitative analyses will be performed to assess the quality of ECG tracings provided by Withings BPM Core and its software, as follows:

* The visibility and polarity of the ECG waves (namely P-waves, QRS complexes and T-waves) will be determined by the cardiologists for each lead I signals recorded with Withings BPM Core and with the 12-channel ECG device. The assessment will be made on the 5th complete beat of the recording. For each of the waves (P, QRS and T), the agreement of visibility and the agreement of polarity (when both are visible) between the signals of Withings BPM Core and the reference ECG device will be computed.
* The duration of the main ECG intervals (namely QT interval, QRS width and PR interval) will be determined by the cardiologists for each lead I signal recorded by Withings BPM Core and the 12-channel ECG device. The measurement will be made with a caliper on the 5th complete beat of the recording. For each interval (QT, QRS, PR), the difference of length between the signals of Withings BPM Core and the reference ECG device will be computed.
* The heart rate will be first determined by the cardiologists for each lead I signal (recorded by Withings BPM Core and the 12-channel ECG device) which are diagnosed as NSR. The heart rate difference between the signals of Withings BPM Core and the reference ECG device will be computed. Second, the heart rate of the signals recorded with the BPM Core will be computed by the Withings software. The difference between the heart rate estimated by Withings software on Withings BPM Core signals and the heart rate determined by the cardiologists on the lead I signal from the ECG reference device will also be calculated.

The sponsor will make sure that the same cardiologist will not be asked to annotate both a Withings BPM Core signal and the corresponding lead I signal from the 12-channel ECG device. The sponsor will then centralize the annotations of Withings BPM Core tracings and of the ECG reference lead I signals and perform agreement calculations on synchronous pairs.

The second secondary objective is to verify the safety of use of the device by analyzing adverse effects.

The safety of use of the device will be assessed by the number of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* male or female who are 18 years or older
* Subject who signed the written informed consent form,
* Able to communicate effectively with and follow instructions from the study staff
* Person with an arm circumference between 22 and 42 cm

Exclusion Criteria:

* Vulnerable subject with regard to regulations

  * Pregnant, parturient or breastfeeding woman,
  * Subject who is deprived of liberty by judicial, medical or administrative decision,
  * Underage subject,
  * Legally protected subject, or subject who is unable to sign the written informed consent form,
  * Subject who is not beneficiary or not affiliated to a social security scheme,
  * Subject within several of the above categories,
* Subject who refused to participate in the study,
* Subject in linguistic or psychic incapacity to sign a written informed consent form,
* Subject in physical incapacity to wear a blood pressure monitor
* Subject with electrical stimulation by pacemaker
* Significant tremor that prevents subject from being able to hold still
* Known sensitivity to medical adhesives, isopropyl alcohol, or ECG electrodes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in and out patients from cardiology services
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the automatic classification in AF by BPM Core single-lead ECG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix AF vs 'non-AF'
Sensitivity of the automatic classification in AF by BPM Core single-lead ECG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix NSR vs 'non-NSR'

SECONDARY OUTCOMES:
Sensitivity of the cardiologists' classification in AF from the BPM Core ECG | 1 year
  sensitivity from the 2x2 confusion matrix AF vs 'non-AF'
Sensitivity of the cardiologists' classification in SR from the BPM Core ECG | 1 year
  sensitivity from the 2x2 confusion matrix NSR vs 'non-NSR'
Accuracy of the visibility of P-waves of single-lead ECG from BPM Core | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the positivity of P-waves of single-lead ECG from BPM Core | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the visibility of QRS-complexes of single-lead ECG from BPM Core | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the positivity of QRS-complexes of single-lead ECG from BPM Core | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the visibility of T-waves of single-lead ECG from BPM Core | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the positivity of T-waves of single-lead ECG from BPM Core | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix

CONTACTS AND LOCATIONS:
Overall Officials: David Campo, PhD, Study Director — Withings
Locations (2):
- France (2):
  - ICPC Floréale, Bagnolet
  - ICPC Turin, Paris

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) are considered as confidential in this study. After the end the final quality control, the database will be frozen and all the IPD will be archived.